CLINICAL TRIAL: NCT00282607
Title: A Randomized, Placebo-Controlled, Double-Blind, Parallel Design Phase 2 Dose Ranging Trial To Assess The Safety and Efficacy of DA-8159 Tablets in Male Subjects With Erectile Dysfunction.
Brief Title: A Study of DA-8159 in Subjects With Erectile Dysfunction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dong-A PharmTech Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DA 2005-001
Record Dates: First submitted 2006-01-25; First posted 2006-01-27 (Estimated); Last update posted 2007-02-28 (Estimated); Status verified 2007-02

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — udenafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: DA-8159

SUMMARY:
The purpose of this study will be to evaluate the clinical efficacy and safety of DA-8159, an orally administered, potent and selective inhibitor of PDE5, versus placebo for the treatment of subjects with erectile dysfunction (ED).

DETAILED DESCRIPTION:
This will be a multi-center, randomized, double-blind, placebo-controlled, parallel-group study in 300 erectile dysfunction patients. Patients will complete a screening visit (V1) to determine eligibility for the study based on the International Index of Erectile Function (IIEF) erectile function (EF) domain scores, patient history and safety measures. Patients that meet the entrance criteria for this study will enter a 4 week, drug-free run-in period to establish a baseline for the erectile function domain score and to meet the criteria for participation in the study.

Patients successfully completing screen will be randomly assigned to one of four treatment groups at Visit 2 (V2): placebo or one of 3 active drug doses of DA-8159 tablets. Patients will be given medication for at-home use and will also be given diaries for recording information regarding sexual encounters, quality of erections and adverse events. At 4-week intervals for 3 months (V3, V4, V5), patients will return to the clinic to review and collect SEP diaries, safety data, 12-lead ECG and medication reconciliation. In addition, at each 4-week interval patients will complete an IIEF, and at Visit 5 will have blood drawn for safety evaluation.

The primary efficacy end points are: a) the change in score (baseline to Visit 5) for the Erectile Function domain score of the IIEF, b) change in response, relative to baseline, for sexual encounter profile (SEP) question 2, and c) change in response, relative to baseline, for SEP question 3. For DA-8159 tablets to be judged efficacious, the DA-8159 tablet groups must be shown superior to the placebo group on all three measures.

ELIGIBILITY:
Inclusion Criteria:

1. Is male and at least 19 years of age.
2. Has a stable monogamous relationship for at least 6 months with a consenting female partner (vaginal intercourse is a required study activity).
3. Provides written informed consent.
4. The subject's female partner provides written informed consent.
5. Has a history of ED (clinically defined as the inability to attain and maintain an erection of the penis sufficient to permit satisfactory sexual intercourse) of at least 3 months duration. The investigator will record the etiology of the ED (organic, psychogenic or mixed).
6. Has scored between 6-25 for the Erectile Function domain score (Questions Number 1-5, 15) at both Visits 1 & 2.
7. Completes least four diary entries by Visit 2, showing at least 4 attempts at sexual intercourse with a 50% or greater failure rate in achieving or in maintaining an erection sufficient to complete intercourse (defined as answering "no" to SEP questions #2 or #3).
8. The subject's partner is not pregnant or lactating and both subject and partner agree to the use of a medically acceptable form of birth control. Exceptions would be subjects with a vasectomy or partners that are post menopausal, and partners that have had a tubal ligation or hysterectomy.

Exclusion Criteria:

1. Has a history of stroke, myocardial infarction, or coronary artery disease within the past 6 months.
2. Has a history of cardiac failure, angina, or life-threatening arrhythmia within the past 6 months.
3. Is taking nitrate medication in any form(Appendix 7)
4. Is taking alpha blockers.
5. Has a clinically significant abnormal laboratory value as determined by the principal investigator.
6. Has a history of uncontrolled diabetes (HbA1c>9%).
7. Has a history of proliferative diabetic retinopathy.
8. Has a history of spinal cord injury or a radical prostatectomy or radical pelvic surgery.
9. Has a supine blood pressure lower than 90/50mmHg or uncontrolled hypertension higher than 170/100mmHg.
10. Has a anatomical deformity of the penis such as severe penile fibrosis or Peyronie's disease.
11. Has a thyroid stimulating hormone (TSH) level lower than 30% of LLN.
12. Has erectile dysfunction caused by neurological or endocrine factors such as hyperprolactinemia or low serum testosterone levels (<300 ng/dl).
13. Has hepatic impairment (GOT, GPT levels > 3 x ULN).
14. Has renal impairment (serum creatinine ≥ 2.5mg/dl).
15. Has a history of hematological disorder such as bleeding disorder or a risk of GI bleeding such as peptic ulceration.
16. Has a history of retinitis pigmentosa.
17. Has a history of sickle cell disease, multiple myeloma, leukemia or any other disorders that may cause priapism.
18. Has a history of significant psychiatric disorder.
19. Has a history of central nervous system disorders such as stroke, transient ischemic attacks, or spinal cord injury.
20. Has a history of drug abuse (alcohol, marijuana, cocaine, or opiates).
21. Has a known sensitivity to drugs especially to phosphodiesterase type 5 inhibitors such as Viagra, Cialis or Levitra.
22. Has used other erectile dysfunction therapies including nutraceutical and herbal products within 14 days prior to entering into this study.
23. Is using concomitant medications that are known or suspected to interact with PDE 5 inhibitors such as the following:

    1. Antibacterial: erythromycin
    2. Antifungals: itraconazole, ketoconazole
    3. Antivirals: ritonavir, saquinavir, amprenavir, indinavir, nelfinavir
    4. H2 receptor antagonist: cimetidine
    5. Anticoagulants, androgens, trazodone
24. Have other sexual disorders such as hypoactive sexual desire.
25. Have previously failed to respond to PDE-5 inhibitors such as Viagra, Cialis or Levitra.
26. Have a major illness that in the opinion of the investigator would interfere with the conduct of the study.
27. Has not participated in a clinical drug study within the last 30 days prior to entering this study.

Ages: 19 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2005-05; Study Completion 2006-06

PRIMARY OUTCOMES:
The primary efficacy end points are:
the change in score (baseline to Visit 5) for the Erectile Function domain score of the IIEF;
change in response, relative to baseline, for sexual encounter profile (SEP) question 2, and
change in response, relative to baseline, for SEP question 3.
Safety will be assessed by monitoring adverse events and changes in vital signs, clinical laboratory test results, 12-lead ECG, and physical examinations.

SECONDARY OUTCOMES:
The study has several secondary efficacy measurements including:
changes in the satisfaction of intercourse, orgasmic function, sexual desire and overall satisfaction domains of the IIEF,
changes from baseline in SEP questions 1, 4 and 5;
the global assessment questionnaire (GAQ), and
changes from baseline in patient self assessment questionnaire (PSAE) scores.

CONTACTS AND LOCATIONS:
Overall Officials: James L Yeager, RPh., Ph.D., Study Director; Harin Padma-Nathan, MD, Principal Investigator — The Male Clinic
Locations (15):
- United States (15):
  - Medical Affiliated Research Center, Huntsville, Alabama
  - The Male Clinic, Beverly Hills, California
  - South Orange County, Laguna Woods, California
  - California Profession Research, Newport Beach, California
  - West Coast Clinical Research, Tarzana, California
  - Urology Research Options, Aurora, Colorado
  - Connecticut Clinical Research Center, Waterbury, Connecticut
  - South Florida Medical Research, Aventura, Florida
  - Florida Foundation for Healthcare Research, Ocala, Florida
  - Northeast Indiana Research, LLC, Fort Wayne, Indiana
  - Drs. Werner, Murdock & Francis, P.A. , Urology Associates, Greenbelt, Maryland
  - Accumed Research Associates, Garden City, New York
  - Center for Urologic Research of Western New York, Williamsville, New York
  - University Urological Researcgh Institute, Providence, Rhode Island
  - Urology San Antonio Research, San Antonio, Texas